CLINICAL TRIAL: NCT04682925
Title: Effect of Evidence-Based Skin Care and Hydrocolloid Dressing in the Prevention of Nasogastric-Related Pressure Injury: A Randomized Controlled Trial
Brief Title: Effect of Evidence-Based Skin Care and Hydrocolloid Dressing in the Prevention of Nasogastric-Related Pressure Injury
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: MAİDE YEŞİLYURT (Other)
Collaborators: Necmettin Erbakan University (Other)
Responsible Party: Sponsor-Investigator, MAİDE YEŞİLYURT, Research Assistant, Necmettin Erbakan University
Organization: Necmettin Erbakan University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: MYesilyurt
Record Dates: First submitted 2020-12-09; First posted 2020-12-24 (Actual); Last update posted 2023-07-21 (Actual); Status verified 2023-07

CONDITIONS: Medical Device Site Injury; Nasogastric Tube; Pressure Injury
Keywords: medical device; medical device-associated pressure injury; nasogastric tube; hydrocolloid dressing; skin care
MeSH Terms: conditions — Pressure Ulcer | interventions — Bandages

STUDY DESIGN:
Intervention Model Description: Prospective Randomized Controlled Clinical Trial
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- skin care arm of where evidence-based practices in the implementation guide (Experimental): Participants in this arm will be given evidence-based skin care interventions, which are included in the guidelines to prevent medical device-related pressure injuries, and are implemented by the researcher nurse. After the nasogastric tube is inserted by the patient's physician.
  Interventions: Other: skin care arm of where evidence-based practices in the implementation guide
- hydrocolloid (Convatec Granuflex-extra thin) dressing (Experimental): Patients in this arm will be applied a translucent hydrocolloid cover, which is compatible with the sensitive skin structure, can be applied to all body surfaces and nasal mucosa, and allows the underlying mucosa and skin to be observed after the nasogastric tube is inserted by the patient's physician. This cover will be applied to the nasal mucosa and nasal wing under the nasogastric tube.
  Interventions: Device: hydrocolloid (Convatec Granuflex-extra thin) dressing
- control (Other): Participants in the control group will be given no intervention , these patients will receive the routine clinical care(dressing change and nasal skin cleaning once a day) applied in the intensive care unit.
  Interventions: Other: control

INTERVENTIONS:
Other: skin care arm of where evidence-based practices in the implementation guide — 1. The nasal mucosa and nasal skin under the nasogastric tube will be cleaned and dried twice a day with a pH-compatible cleanser.
  2. A water-based moisturizing cream will be applied to the nasal skin under the nasogastric tube twice a day, after care with a pH-compatible cleanser.
  3. Spray skin barrier will be applied twice a day after applying water-based moisturizing cream to the nasal skin under the nasogastric tube.
  4. The nasal mucosa and nasal skin under the nasogastric tube will be evaluated twice daily for signs of pressure-related injury. All these care interventions applied to the skin care arm will be applied together with the doctor and nurse responsible for the treatment and care of the patient.
  Arms: skin care arm of where evidence-based practices in the implementation guide
Device: hydrocolloid (Convatec Granuflex-extra thin) dressing — The nasal skin of the patients and the surrounding skin will be cleaned with a pH-compatible cleaner, dried and a new hydrocolloid cover will be applied once a day. All these care interventions applied to the hydrocolloid dressing arm will be applied together with the physician and nurse responsible for the treatment and care of the patient.
  Arms: hydrocolloid (Convatec Granuflex-extra thin) dressing
Other: control — In routine care, the skin under the nasogastric tube is evaluated once a day for redness and wound formation by the nurse responsible for the patient's care and is cleaned and dried with appropriate cleaners.
  Arms: control

SUMMARY:
This study was planned as a prospective randomized controlled clinical trial to determine the effect of evidence-based skin care interventions and hydrocolloid dressings in preventing nasogastric induced pressure injuries in critically ill patients.

DETAILED DESCRIPTION:
Intensive care patients in whom a large number of medical devices are applied during the treatment and care process are at risk for medical device-related pressure injuries.One of the most common medical tools applied to these patients is the nasogastric tube.These tubes, which are applied to provide nasal decompression and enteral nutrition, cause pressure injuries in the nasal mucosa and nasal wings of the patients.These wounds prevent the patient from feeding, delay the healing process by causing the nasogastric tube to be pulled, delay the healing process, cause the patient to experience discomfort and pain by re-inserting the tube from the other nostril, and increase the cost of treatment and care.Guidelines for prevention of pressure injuries, which include evidence-based recommendations, report that these wounds can be prevented with evidence-based skin care interventions and hydrocolloid dressings. This study was planned as a prospective randomized controlled clinical trial to determine the effect of evidence-based skin care interventions and hydrocolloid dressings in preventing nasogastric induced pressure injuries in critically ill patients. In the literature, there is no study evaluating the effect of evidence-based skin care and / or hydrocolloid dressings on pressure injuries caused by nasogastric tube. Therefore, a study demonstrating that hydrocolloid dressing reduce pressure injuries to the nasal arch due to non-invasive mechanical ventilation were referenced in the sample calculation. In the sample selection, it was determined that the rate of pressure injury (n: 27/49) developed more in those who did not use hydrocolloids than those who were used (n: 6/73). In the sample calculation made in the G * Power (3.1.9.2) program, it was determined that a total of 56 patients, including at least 28 patients in each study group, should be included in the sample. It was predicted that 20% of the sample could be lost during the data collection process, and in this study, which was planned with three arms (control, skin care, hydrocolloid dressing), it was determined that the research sample should be 102, with at least 34 patients on each arm. The patients included in the study will be assigned to the experimental group (skin care, hydrocolloid dressing) and control group by balanced block randomization method according to the randomization list in a ratio of 1: 1:1. In the study, block randomization was performed by a statistician based on the patients age. The final evaluation of the patients included in the study will be made on the day of the wound in those with pressure sores. In other patients, it will be performed on the 18th day of the nasogastric tube, considering the literature data that pressure injuries occur within 2-7 and 11 ± 6.17 days after tube insertion. For those whose nasogastric tube is removed before the 18th day, the last follow-up will be done on the day the tube is removed. For the implementation of the study, permission was obtained from the ethics committee of Republic of Turkey Ministry of Health, Turkey Pharmaceuticals and Medical Devices Agency Ethics Committee, and work permit was obtained from Necmettin Erbakan University Meram Medical Faculty Hospital Chief Physician. Patients/patient guardian included in the study sample will be informed before the study that the purpose of the study and participation in the study is in line with the principle of volunteering, and "Informing and Consent of Volunteers Consent Form" will be signed.

Data collection tools;

* Personal Information Form,
* The form containing the characteristics of the treatment and care process in the Intensive Care Unit
* The form containing the features associated with the nasogastric tube,
* A chart recording the state of nasogastric tube pressure injury, the area of occurrence and its stage, Independent variables
* Identifying features of patients,
* Evaluations and follow-ups during the treatment and care process,
* Interventions to prevent nasogastric tube pressure injury (routine clinical care, evidence-based skin care interventions, hydrocolloid dressing) Dependent variables
* Pressure injury originating from nasogastric tube Evaluation of the Data In the evaluation of the descriptive data obtained from the research, number, percentage, average and standard deviation will be used; The conformity of the data to normal distribution will be determined by Kolmogorov-Smirnov test and normal distribution curve, Skewness and Kurtosis test, and when the data show normal distribution, parametric tests will be used, and nonparametric tests will be used in the analysis of data that do not conform to the normal distribution. Significance will be evaluated within the confidence interval of 95%, p <0.05 will be taken.

İmplementation of the research Patients who are 18 years of age or older, who have a nasogastric tube inserted after admission to the intensive care unit, and whose nasogastric tube stay is planned to be at least 48 hours will be included in the sample group.

Participants in the experimental group( evidence-based skin care), evidence-based skin care interventions in the guidelines to prevent medical device-related pressure injuries will be applied twice daily to the nasal mucosa and nasal wing under the nasogastric tube.

Participants in the experimental group( hydrocolloid dressing), hydrocolloid dressing will be applied daily to the nasal mucosa and nasal wing of the patients under the nasogastric tube to prevent pressure injuries caused by medical devices.

Participants in the control group will be given no intervention , these patients will receive the routine care(dressing change and nasal skin cleaning once a day) applied in the intensive care unit.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older,
* Having written permission from relatives and / or him / her,
* A nasogastric tube is inserted after admission to the Intensive Care Unit,
* In accordance with the literature reporting that nasogastric tube-induced pressure injuries occur on the second day after nasogastric tube, patients with a planned nasogastric tube stay of at least 48 hours will be included.

Exclusion Criteria:

* Do not sign the informed consent form,
* A nasogastric tube inserted during admission to the Intensive Care Unit,
* If there is irritation or wound in the nasal mucosa, nasal arch, nasal wings and surrounding tissue before the nasogastric tube is inserted,
* A rash that does not fade with pressure on the nasal arch, nose wings and surrounding tissue before the nasogastric tube is inserted,
* Nasogastric tube position change is contraindicated.
* Nasal intubation is applied before the nasogastric tube is inserted,
* If nasogastric tube stay is planned to be shorter than 48 hours, patients will not be included.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 102 (Actual)
Dates: Start 2021-01-15 (Actual); Primary Completion 2022-01-15 (Actual); Study Completion 2022-06-15 (Actual)

PRIMARY OUTCOMES:
rate of pressure injury from nasogastric tube | Each participant will be followed for 18 days
  Pressure injury originating from nasogastric tube will be evaluated with the reliable international NPUAP / EPUAP Pressure Ulcer Classification System. In the literature, pressure injuries originating from nasogastric tube are reported to develop in 11± 5 days. Accordingly, patients will be cared for and followed up for 18 days. The day the pressure injury develops will be recorded in each group.

SECONDARY OUTCOMES:
The most effective intervention in preventing pressure injuries caused by nasogastric tube | Each participant will be followed for 18 days
  It recommends evidence-based practices, twice-daily skin care or daily prophylactic dressing to prevent nasogastric tube-induced pressure injuries. The most effective method to prevent pressure injury will be revealed. Pressure injury originating from nasogastric tube will be evaluated with the reliable international NPUAP / EPUAP Pressure Ulcer Classification System.

CONTACTS AND LOCATIONS:
Overall Officials: SERPİL YÜKSEL, PhD, Principal Investigator — Necmettin Erbakan University; ALPER YOSUNKAYA, PhD, Study Director — Necmettin Erbakan University; MAİDE YEŞİLYURT, MSc, Study Director — Necmettin Erbakan University
Locations (1):
- Necmettin Erbakan University, Konya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
STUDY PROTOCOL
Supporting Information: Study Protocol

REFERENCES:
- [Derived] Yesilyurt M, Yuksel S, Yosunkaya A. The effect of evidence-based skin care and hydrocolloid dressing in the prevention of nasogastric tube-related pressure injury: A randomized controlled clinical trial. J Tissue Viability. 2024 Nov;33(4):889-894. doi: 10.1016/j.jtv.2024.09.001. Epub 2024 Sep 12. PMID 39289093